CLINICAL TRIAL: NCT02947789
Title: Predictive Model for Postoperative Mortality in Adult Emergency Surgical Patients Under General Anesthesia
Brief Title: Predictive Model for Postoperative Mortality
Status: Completed | Type: Observational
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Thepakorn Sathitkarnmanee, Associate Professor, Khon Kaen University
Other Study IDs: HE581131
Record Dates: First submitted 2016-10-26; First posted 2016-10-28 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Postoperative Complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Postoperative mortality within 3 days: Group 1: Patients undergoing emergency surgery with postoperative mortality within 3 days Group 2: Patients undergoing emergency surgery without postoperative mortality within 3 days
  Interventions: Procedure: Emergency surgery

INTERVENTIONS:
Procedure: Emergency surgery — Patients undergoing emergency surgery

SUMMARY:
Surgery has risk of morbidity and mortality. Risk factors include: patient factors; surgical factors; and anesthetic factors. The risk is much higher in emergency cases. The study of relevant risk factors can lead to improvement in patient management and reduction in mortality.

DETAILED DESCRIPTION:
Objective: To identify risk factors for postoperative mortality within 3 days in adult patients undergoing emergency surgery and construct a predictive model.

Methods: This will be a retrospective, exploratory and analytical study. All medical records of adult patients undergoing emergency surgery between January 2013 to December 2014 will be used to analyze for relevant risk factors using binary logistic regression analysis. A predictive model to predict postoperative morbidity within 3 days will be constructed.

ELIGIBILITY:
Inclusion Criteria:

* Emergency surgery
* Age => 18 years

Exclusion Criteria:

* Caesarean section
* Incomplete medical record

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing emergency surgery
Sampling Method: Non-Probability Sample
Enrollment: 740 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Postoperative mortality within 3 days | through study completion, an average of 1 week
  Patient die postoperatively within 3 day3

CONTACTS AND LOCATIONS:
Overall Officials: Sirirat Tribuddharat, MD, Principal Investigator — Faculty of Medicine, Khon Kaen University, Khon Kaen, Thailand
Locations (1):
- Faculty of Medicine, Khon Kaen University, Khon Kaen, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Akinbami F, Askari R, Steinberg J, Panizales M, Rogers SO Jr. Factors affecting morbidity in emergency general surgery. Am J Surg. 2011 Apr;201(4):456-62. doi: 10.1016/j.amjsurg.2010.11.007. PMID 21421099
- [Result] Fukuda N, Wada J, Niki M, Sugiyama Y, Mushiake H. Factors predicting mortality in emergency abdominal surgery in the elderly. World J Emerg Surg. 2012 May 11;7(1):12. doi: 10.1186/1749-7922-7-12. PMID 22578159
- [Result] Ingraham AM, Cohen ME, Bilimoria KY, Raval MV, Ko CY, Nathens AB, Hall BL. Comparison of 30-day outcomes after emergency general surgery procedures: potential for targeted improvement. Surgery. 2010 Aug;148(2):217-38. doi: 10.1016/j.surg.2010.05.009. PMID 20633727
- [Result] Matsuyama T, Iranami H, Fujii K, Inoue M, Nakagawa R, Kawashima K. Risk factors for postoperative mortality and morbidities in emergency surgeries. J Anesth. 2013 Dec;27(6):838-43. doi: 10.1007/s00540-013-1639-z. Epub 2013 May 23. PMID 23700220
- [Result] Wilson I, Paul Barrett M, Sinha A, Chan S. Predictors of in-hospital mortality amongst octogenarians undergoing emergency general surgery: a retrospective cohort study. Int J Surg. 2014 Nov;12(11):1157-61. doi: 10.1016/j.ijsu.2014.08.404. Epub 2014 Sep 16. PMID 25229887